CLINICAL TRIAL: NCT01373515
Title: Phase 1 Study of Leukemic Dendritic Cell Vaccination in Patients With Acute Myeloid Leukemia
Brief Title: Leukemic Dendritic Cell Vaccination in Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mendus (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DCOne-1
Record Dates: First submitted 2011-05-30; First posted 2011-06-15 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Acute Myeloid Leukemia (AML); Leukemic Dendritic Cell Vaccination
Keywords: DCOne; DCP-001; Second complete remission of AML; Relapse AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1; 1x10E7 DCP-001 (Experimental): n=3; patients receiving 4 bi-weekly vaccinations of 1x10E7 DCP-001.
  Interventions: Biological: DCP-001
- Cohort 2; 2.5x10E7 DCP-001 (Experimental): n=3; patients receiving 4 bi-weekly vaccinations of 2.5x10E7 DCP-001.
  Interventions: Biological: DCP-001
- Cohort 3; 5x10E7 DCP-001 (Experimental): n=3; patients receiving 4 bi-weekly vaccinations of 5x10E7 DCP-001.
  Interventions: Biological: DCP-001
- Cohort 4; 5x10E7 DCP-001 (Experimental): n=3; patients, matched for HLA-A2, receiving 4 bi-weekly vaccinations of 5x10E7 DCP-001. Or, in case this turned out toxic, this group will receive the Maximum Tolerated Dose.
  Interventions: Biological: DCP-001

INTERVENTIONS:
Biological: DCP-001 — 4 bi-weekly vaccinations

SUMMARY:
This is an open label phase 1 feasibility and safety dose escalation study. The main objective is to evaluate the safety of DCP-001 intradermal vaccination in patients with AML.

DETAILED DESCRIPTION:
DCPrime is testing an allogeneic (non-self cells, standardised product) DC-based immunotherapy in cancer patients. The technology consists of sustainable dendritic progenitor cells (named "DCOne™") and a proprietary method to expand these and to create functional mature dendritic cells (DCP-001).

AML is a fast growing form of leukemia that particularly in the elderly (>60) is life threatening. As age is an important factor in determining the success of AML treatment, overall, AML has a bad prognosis as only 24% of the patients are alive 5 years after diagnosis.

Without treatment AML is fatal, usually within months. Chemotherapy can cure patients and prolong survival in responders; however, chemotherapy is also quite toxic and can cause substantial morbidity and mortality. The most commonly prescribed first line therapy for patients with AML is a combination of an anthracycline and cytarabine; in the Western world the anthracycline is either daunorubicin or idarubicin. Post remission therapy (consolidation therapy) is usually given.

There is therefore substantial medical need for new treatment modalities. One of the major difficulties regarding development of new agents is that relatively low response rates and toxicity issues have been in the way of approval of new agents. Immunotherapy, in particular with the therapeutic vaccines, is expected to have potential in prevention of recurrence of disease after cytoreductive therapy. Any drug that could prevent or reduce minimal residual disease in the population is likely to meet a strong medical need for this population of high risk patients.

In this phase 1 trial consecutive eligible patients will be treated until 12 patients have completed the study. Patients will be started with the vaccination program within 2 months after having achieved complete remission or in patients who have stable disease over at least a 2 month period.

The first cohort (n=3) will receive 4 bi-weekly vaccinations of 1x10E7 DCP-001, the second cohort (n=3) will receive 4 bi-weekly vaccinations of 2.5x10E7 DCP-001, and the last cohort (n=3) will receive 4 bi-weekly vaccinations of 5x10E7 DCP-001. The Dose Limiting Toxicity (DTL) is defined as non-hematological toxicity of ≥ 3 according to common toxicity criteria v3.0. The 4th cohort (matched for HLA-A2) will receive 4 vaccinations of the highest dose (5x10E7 DCP-001) or, in case this turned out to be toxic (as determined by the vaccination profile of cohort 1, 2 and 3), this group will receive the Maximum Tolerated Dose (MTD).

DCP-001 vaccine is presented as a direct injectable sterile cell suspension consisting of irradiated mature dendritic cells in cryopreservation solution packed in vials. The vaccine will be administered intradermally.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML, in second complete remission of AML (all FAB-subclasses), not eligible for additional intensification therapies e.g. allogeneic (allo) PSCT [independent of age]; OR
* Patients with relapse (smouldering) AML not eligible for additional intensification therapies e.g. alloPSCT; OR
* Patients with de novo (smouldering) AML not eligible for intensive treatment according to current HOVON trials.
* Patients >65 years of age with de novo AML in first CR and off protocol of current HOVON trials.
* WHO performance of 0, 1, or 2.
* Male or female patients at least 18 years of age and <80 years by date of enrolment.
* Patients not treated within current HOVON or other AML trials.
* Ability and willingness to give informed consent.
* HLA-A2.1 positive patients (only for cohort 4).

Exclusion Criteria:

* Uncontrolled active infection.
* Previous immunotherapy in last 3 months (except for anti-CD33 targeted therapy).
* Previous allogeneic PSCT.
* Inadequate bone marrow function: absolute neutrophile count (ANC) < 0.5x10E9/L, or platelet count < 20x10E9/L or active bleeding with platelet count > 20x10E9/L.
* Inadequate liver function, defined as:

  * Serum (total) bilirubin > 1.5 x the upper limit of normal (ULN)
  * AST/SGOT or ALT/SGPT > 2.5 x ULN
  * Alkaline phosphatase levels > 2.5 times the ULN at baseline.
* Inadequate renal function, defined as:

  * Serum creatinine > 1.5 x ULN
* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
* Pregnant or lactating females. Serum pregnancy test to be assessed within 7 days prior to study treatment start, or within 14 days with a confirmatory urine pregnancy test within 7 days prior to study treatment start.
* Women of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) not using effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly).
* Major surgical procedure (including open biopsy) within 28 days prior to the first study treatment, or anticipation of the need for major surgery during the course of the study treatment.
* Minor surgical procedures, within 24 hours prior to the first study treatment.
* Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident (CVA) / stroke within ≤ 6 months prior to the first study treatment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia requiring medication.
* Known hypersensitivity to any of the study drugs or excipients.
* Evidence of an other medical condition (such as psychiatric illness, physical examination or laboratory findings that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.
* Eligibility for the HOVON-93 study (intensification program ± allogeneic stem cell transplant).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety/Feasibility of DCP-001 vaccination | three months and follow up after study completion
  The primary endpoint of this study will be the safety and feasibility of DCP-001 vaccination in AML patients. Safety will be assessed by means of laboratory evalulations, lhysical examination, vital sign assessments and adverse events recording. Clinical efficacy is assessed by the presence of leukemic cells in blood and bonemarrow and physical examination at baseline, during and after vaccination

SECONDARY OUTCOMES:
Immunological responses induced by DCP-001 vaccination | 3 months
  The secondary endpoint of this study will be establishment of immunological responses induced by DCP-001 vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands